CLINICAL TRIAL: NCT01335399
Title: A Phase 3, Randomized, Open Label Trial of Lenalidomide/Dexamethasone With or Without Elotuzumab in Subjects With Previously Untreated Multiple Myeloma
Brief Title: Phase III Study of Lenalidomide and Dexamethasone With or Without Elotuzumab to Treat Newly Diagnosed, Previously Untreated Multiple Myeloma
Acronym: ELOQUENT - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-006; 2010-022445-20 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed; Previously Untreated
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide + Dexamethasone (Active Comparator)
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- Lenalidomide + Dexamethasone + Elotuzumab (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Biological: Elotuzumab (BMS-901608; HuLuc63)

INTERVENTIONS:
Drug: Lenalidomide — Capsules, Oral, 25 mg, once daily, on Days 1-21, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Revlimid®
Drug: Dexamethasone — Tablets, Oral, 40 mg, weekly, on Days 1, 8, 15, 22, Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone
Drug: Dexamethasone — Tablets, Oral, 28 mg, once daily, on Days 1, 8, 15, 22 (cycles 1&2) ; Days 1 &15 (cycles 3-18); Day 1 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone + Elotuzumab
Drug: Dexamethasone — Tablets, Oral, 40 mg, once daily, on Days 8 & 22 (cycles 3-18); Days 8, 15, 22 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone + Elotuzumab
Drug: Dexamethasone — Solution, Intravenous (IV), 8 mg, Once daily, on Days 1, 8, 15, 22 (cycles 1&2) ; Days 1 &15 (cycles 3-18); Day 1 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
  Arms: Lenalidomide + Dexamethasone + Elotuzumab
Biological: Elotuzumab (BMS-901608; HuLuc63) — Solution, Intravenous (IV), 10 mg/kg, weekly, on Days 1, 8, 15, 22 (cycles 1&2); Days 1 and 15 (cycles 3-18), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Arms: Lenalidomide + Dexamethasone + Elotuzumab
Biological: Elotuzumab (BMS-901608; HuLuc63) — Solution, Intravenous (IV), 20 mg/kg, Day 1 (cycle 19 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Arms: Lenalidomide + Dexamethasone + Elotuzumab

SUMMARY:
The purpose of the study is to determine whether the addition of Elotuzumab to Lenalidomide/low-dose Dexamethasone will increase the progression free survival (PFS)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects who are newly diagnosed with symptomatic Multiple Myeloma (MM) and who:

  * have not received any prior systemic anti-myeloma therapy AND
  * have measurable disease AND
  * are not candidates for high-dose therapy plus stem-cell transplantation (SCT) because of age (≥ 65 years) or coexisting conditions. Refusal to undergo high dose therapy with SCT is NOT sufficient for entry onto CA204006 for a subject < 65 years old. There must be a comorbidity that prevents SCT for a subject < 65 years old

Exclusion Criteria:

* Subjects with non-secretory or oligo-secretory or free light-chain only myeloma
* Smoldering MM, defined as asymptomatic MM with absence of lytic bone lesions
* Monoclonal Gammopathy of Undetermined Significance (MGUS)
* Active plasma cell leukemia
* Known Human Immunodeficiency Virus (HIV) infection or active hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2011-08-04 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (235):
- United States (88):
  - Local Institution - 1628, Birmingham, Alabama
  - Local Institution - 7619, Mobile, Alabama
  - Local Institution - 7618, Mobile, Alabama
  - Local Institution - 7617, Chandler, Arizona
  - Local Institution - 1644, Tucson, Arizona
  - Local Institution - 1618, Bakersfield, California
  - Local Institution - 1602, Berkeley, California
  - Local Institution - 1636, Corona, California
  - Local Institution - 1668, Corona, California
  - Local Institution - 1616, Greenbrae, California
  - Local Institution - 7609, Long Beach, California
  - Local Institution - 1660, Los Angeles, California
  - Local Institution - 1673, Orange, California
  - Local Institution - 1613, San Diego, California
  - Local Institution - 1621, New Haven, Connecticut
  - Local Institution - 1612, Washington D.C., District of Columbia
  - Local Institution - 1682, Boca Raton, Florida
  - Local Institution - 1617, Brooksville, Florida
  - Local Institution - 1648, Fort Myers, Florida
  - Local Institution - 7613, Hollywood, Florida
  - Local Institution - 1623, Jacksonville, Florida
  - Local Institution - 1625, New Port Richey, Florida
  - Local Institution - 1649, St. Petersburg, Florida
  - Local Institution - 1611, West Palm Beach, Florida
  - Local Institution - 1630, Atlanta, Georgia
  - Local Institution - 1684, Honolulu, Hawaii
  - Local Institution - 1607, Chicago, Illinois
  - Local Institution - 1635, Chicago, Illinois
  - Local Institution - 1632, Maywood, Illinois
  - Local Institution - 7606, Peoria, Illinois
  - Local Institution - 7610, Skokie, Illinois
  - Local Institution - 1603, Urbana, Illinois
  - Local Institution - 7616, Bloomington, Indiana
  - Local Institution - 7620, Indianapolis, Indiana
  - Local Institution - 1669, Indianapolis, Indiana
  - Local Institution - 1656, Mishawaka, Indiana
  - Local Institution - 1633, Iowa City, Iowa
  - Local Institution - 1674, Lexington, Kentucky
  - Local Institution - 1683, Louisville, Kentucky
  - Local Institution - 1646, Lafayette, Louisiana
  - Local Institution - 7614, Marrero, Louisiana
  - Local Institution - 1626, New Orleans, Louisiana
  - Local Institution - 1652, Shreveport, Louisiana
  - Local Institution - 1676, Baltimore, Maryland
  - Local Institution - 1650, Baltimore, Maryland
  - Local Institution - 1619, Boston, Massachusetts
  - Local Institution - 1699, Boston, Massachusetts
  - Local Institution - 1604, Detroit, Michigan
  - Local Institution - 1667, Jefferson City, Missouri
  - Local Institution - 1651, Springfield, Missouri
  - Local Institution - 1645, St Louis, Missouri
  - Local Institution - 1637, Omaha, Nebraska
  - Local Institution - 7621, Mineola, New York
  - Local Institution - 1615, New York, New York
  - Local Institution - 1671, Stony Brook, New York
  - Local Institution - 7604, Goldsboro, North Carolina
  - Local Institution - 1610, Winston-Salem, North Carolina
  - Local Institution - 1608, Cleveland, Ohio
  - Local Institution - 1693, Cleveland, Ohio
  - Local Institution - 1638, Columbus, Ohio
  - Local Institution - 1664, Columbus, Ohio
  - Local Institution - 1690, Middletown, Ohio
  - Local Institution - 1655, Tulsa, Oklahoma
  - Local Institution - 7611, Langhorne, Pennsylvania
  - Local Institution - 1647, Pittsburgh, Pennsylvania
  - Local Institution - 1679, Pittsburgh, Pennsylvania
  - Local Institution - 1677, Sayre, Pennsylvania
  - Local Institution - 1629, Charleston, South Carolina
  - Local Institution - 7615, Charleston, South Carolina
  - Local Institution - 1624, Greenville, South Carolina
  - Local Institution - 7607, Sioux Falls, South Dakota
  - Local Institution - 1600, Knoxville, Tennessee
  - Local Institution - 7628, Memphis, Tennessee
  - Local Institution - 1627, Nashville, Tennessee
  - Local Institution - 1670, Nashville, Tennessee
  - Local Institution - 1634, Corpus Christi, Texas
  - Local Institution - 7612, Dallas, Texas
  - Local Institution - 1643, Houston, Texas
  - Local Institution - 1686, Houston, Texas
  - Local Institution - 1642, Houston, Texas
  - Local Institution - 7623, Ogden, Utah
  - Local Institution - 1657, Fredericksburg, Virginia
  - Local Institution - 1640, Seattle, Washington
  - Local Institution - 1631, Seattle, Washington
  - Local Institution - 1601, Huntington, West Virginia
  - Gundersen Clinic, Ltd, La Crosse, Wisconsin
  - Local Institution - 1663, Madison, Wisconsin
  - Local Institution - 1609, Madison, Wisconsin
- Australia (13):
  - Local Institution - 3600, Garran, Australian Capital Territory
  - Local Institution - 3607, Waratah, New South Wales
  - Local Institution - 3610, Westmead, New South Wales
  - Local Institution - 3609, Herston, Queensland
  - Local Institution - 3608, Milton, Queensland
  - Local Institution - 3612, Adelaide, South Australia
  - Local Institution - 3606, Woodville South, South Australia
  - Local Institution - 3601, Fitzroy, Victoria
  - Local Institution - 3602, Frankston, Victoria
  - Local Institution - 3603, Heidelberg Melbourne, Victoria
  - Local Institution - 3604, Wodonga, Victoria
  - Local Institution - 3605, Murdoch
  - Local Institution - 3611, Nedlands
- Austria (4):
  - Local Institution - 4052, Fadingerstraße 1
  - Local Institution - 4051, Innsbruck
  - Local Institution - 4054, Rankweil
  - Local Institution - 4053, Wels
- Belgium (9):
  - Local Institution - 4160, Brussels
  - Local Institution - 4156, Brussels
  - Local Institution - 4157, Brussles
  - Local Institution - 4154, Charleroi
  - Local Institution - 4159, Haine-Saint-Paul
  - Local Institution - 4158, Leuven
  - Local Institution - 4150, Liège
  - Local Institution - 4153, Roeselare
  - Local Institution - 4151, Yvoir
- Canada (10):
  - Local Institution - 2601, Calgary, Alberta
  - Local Institution - 2600, Edmonton, Alberta
  - Local Institution - 2602, Winnipeg, Manitoba
  - Local Institution - 2611, Saint John, New Brunswick
  - Local Institution - 2610, Halifax, Nova Scotia
  - Local Institution - 2606, London, Ontario
  - Local Institution - 2612, Toronto, Ontario
  - Local Institution - 2603, Greenfield Park, Quebec
  - Local Institution - 2605, Montreal, Quebec
  - Local Institution - 2607, Montreal, Quebec
- Czechia (3):
  - Local Institution - 4252, Hradec Králové
  - Local Institution - 4250, Prague
  - Local Institution - 4251, Prague
- Germany (15):
  - Local Institution - 4565, Aschaffenburg
  - Local Institution - 4550, Berlin
  - Local Institution - 4555, Chemnitz
  - Local Institution - 4563, Cologne
  - Local Institution - 4562, Dresden
  - Local Institution - 4552, Hamm
  - Local Institution - 4553, Heidelberg
  - Local Institution - 4560, Jena
  - Local Institution - 4554, Mainz
  - Local Institution - 4561, München
  - Local Institution - 4558, Münster
  - Local Institution - 4551, Offenbach
  - Local Institution - 4556, Stuttgart
  - Local Institution - 4564, Tübingen
  - Local Institution - 4559, Ulm
- Greece (5):
  - Local Institution - 4653, Athens
  - Local Institution - 4651, Athens
  - Local Institution - 4650, Ioannina
  - Local Institution - 4652, Larissa
  - Local Institution - 4654, Pátrai
- Hungary (5):
  - Local Institution - 4751, Budapest
  - Local Institution - 4754, Budapest
  - Local Institution - 4750, Debrecen
  - Local Institution - 4753, Győr
  - Local Institution - 4752, Szeged
- Ireland (3):
  - Local Institution - 4852, Dublin
  - Local Institution - 4850, Dublin
  - Local Institution - 4851, Galway
- Israel (10):
  - Local Institution - 4950, Afula
  - Local Institution - 4956, Ashkelon
  - Local Institution - 4960, Haifa
  - Local Institution - 4958, Jerusalem
  - Local Institution - 4951, Jerusalem
  - Local Institution - 4959, Kfar Saba
  - Local Institution - 4954, Nahariya
  - Local Institution - 4952, Petah Tikva
  - Local Institution - 4957, Tel Aviv
  - Local Institution - 4955, Ẕerifin
- Italy (21):
  - Local Institution - 5067, Ancona
  - Local Institution - 5065, Bari
  - Local Institution - 5053, Bergamo
  - Local Institution - 5070, Bologna
  - Local Institution - 5066, Florence
  - Local Institution - 5050, Genova
  - Local Institution - 5057, Meldola
  - Local Institution - 5069, Milan
  - Local Institution - 5075, Milan
  - Local Institution - 5052, Monza
  - Local Institution - 5062, Napoli
  - Local Institution - 5068, Napoli
  - Local Institution - 5055, Palermo
  - Local Institution - 5063, Ravenna
  - Local Institution - 5073, Reggio Nell Emilia (RE)
  - Local Institution - 5064, Rimini
  - Local Institution - 5058, Roma
  - Local Institution - 5054, Roma
  - Local Institution - 5056, Rome
  - Local Institution - 5072, Terni
  - Local Institution - 5051, Torino
- Poland (12):
  - Local Institution - 5250, Bialystok
  - Local Institution - 5252, Chorzów
  - Local Institution - 5254, Gdansk
  - Local Institution - 7626, Krakow
  - Local Institution - 5258, Lodz
  - Local Institution - 5257, Lublin
  - Local Institution - 5259, Poznan
  - Local Institution - 5255, Szczecin
  - Local Institution - 5256, Warsaw
  - Local Institution - 5253, Warsaw
  - Local Institution - 5260, Warsaw
  - Local Institution - 5251, Wroclaw
- Puerto Rico (2):
  - Local Institution - 7600, Ponce
  - Local Institution - 7602, San Juan
- Romania (6):
  - Local Institution - 5356, Brasov
  - Local Institution - 5350, Bucaresti
  - Local Institution - 5355, Bucharest
  - Local Institution - 5353, Bucharest
  - Local Institution - 5352, Bucharest
  - Local Institution - 5351, Lasi
- Russia (3):
  - Local Institution - 5450, Saint Petersburg
  - Local Institution - 5452, Saint Petersburg
  - Local Institution - 5453, Samara
- Spain (12):
  - Local Institution - 5552, Badalona-barcelona
  - Local Institution - 5559, Barcelona
  - Local Institution - 5555, Barcelona
  - Local Institution - 5557, Donostia / San Sebastian
  - Local Institution - 5561, La Laguna- Tenerife
  - Local Institution - 5553, Madrid
  - Local Institution - 5551, Madrid
  - Local Institution - 5560, Madrid
  - Local Institution - 5554, Madrid
  - Local Institution - 5558, Pamplona
  - Local Institution - 5550, Salamanca
  - Local Institution - 5556, Toledo
- Switzerland (4):
  - Local Institution - 5751, Bern
  - Local Institution - 5750, Sankt Gallen
  - Local Institution - 5753, Zurich
  - Local Institution - 5752, Zurich
- Turkey (Türkiye) (4):
  - Local Institution - 5853, Izmir, Bornova
  - Local Institution - 5851, Ankara, Dikimevi
  - Local Institution - 5854, Izmir, Inciralti
  - Local Institution - 5856, Gaziantep
- United Kingdom (6):
  - Local Institution - 5951, Belfast, Antrim
  - Local Institution - 5953, London, Greater London
  - Local Institution - 5950, London
  - Local Institution - 5954, London
  - Local Institution - 5952, London
  - Local Institution - 5955, London

REFERENCES:
- [Derived] Dimopoulos MA, Richardson PG, Bahlis NJ, Grosicki S, Cavo M, Beksac M, Legiec W, Liberati AM, Goldschmidt H, Belch A, Magen H, Larocca A, Laubach JP, Petrucci MT, Reece D, White D, Mateos MV, Spicka I, Lazaroiu M, Berdeja J, Kaufman JL, Jou YM, Ganetsky A, Popa McKiver M, Lonial S, Weisel K; ELOQUENT-1 investigators. Addition of elotuzumab to lenalidomide and dexamethasone for patients with newly diagnosed, transplantation ineligible multiple myeloma (ELOQUENT-1): an open-label, multicentre, randomised, phase 3 trial. Lancet Haematol. 2022 Jun;9(6):e403-e414. doi: 10.1016/S2352-3026(22)00103-X. Epub 2022 May 9. PMID 35550060
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- E-Ld Cohort: Participants receiving a combination of Elotuzumab (E) Lenalidomide (L) Dexamethasone (d) in a 28 day cycle
- Ld Cohort: Participants receiving a combination of Lenalidomide (L) Dexamethasone (d) in a 28 day cycle
Period: Pre-treatment Period
Arm/Group | E-Ld Cohort | Ld Cohort
Started (Started = randomized) | 374 | 374
Completed (Completed = continued to the treatment period) | 371 | 371
Not Completed | 3 | 3
Not completed — No longer meeting study criteria | 0 | 1
Not completed — Participant request to discontinue | 0 | 1
Not completed — Adverse event unrelated to study drug | 0 | 1
Not completed — Consent withdrawal | 3 | 0
Period: Treatment Period
Arm/Group | E-Ld Cohort | Ld Cohort
Started | 371 | 371
Completed | 0 | 0
Not Completed | 371 | 371
Not completed — Disease progression | 117 | 145
Not completed — Adverse event unrelated to study drug | 110 | 73
Not completed — Study drug toxicity | 52 | 64
Not completed — Participant request to discontinue | 30 | 22
Not completed — Other reasons | 30 | 30
Not completed — Consent withdrawal | 10 | 7
Not completed — Death | 7 | 6
Not completed — Poor/Non-compliance | 3 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Maximum clinical benefit | 1 | 1
Not completed — No longer meet study criteria | 1 | 1
Not completed — Administrative reasons by Sponsor | 8 | 16

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Ld Cohort | Ld Cohort | Total
Number analyzed (Participants) | 374 | 374 | 748
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.9 (6.58) | 73.1 (6.70) | 73.0 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 173 | 336
  Male | 211 | 201 | 412
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 70 | 87 | 157
  Unknown or Not Reported | 295 | 279 | 574
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 16 | 29
  White | 360 | 351 | 711
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of the first documented tumor progression (as determined by the Independent Review Committee (IRC)) or death due to any cause.
  The IRC conducted a blinded, independent review of the tumor assessments based on the European Group for Blood and Bone Marrow Transplant (EBMT) criteria.
  Censoring rules applied:
  * Participants receiving subsequent systemic anti-myeloma therapy prior to documented progression were censored at the date of the last adequate tumor assessment prior to new therapy.
  * Participants who had an event (progression or death) > 10 weeks after their last tumor assessment were censored at their last adequate tumor assessment prior to the event.
  * Participants without progression or death (and not receiving subsequent therapy prior to progression) were censored at their last adequate tumor assessment.
  * Participants without any post-baseline tumor assessments were censored on the date of randomization
Time Frame: From randomization to date of first documented tumor progression or death due to any cause (up to 8 years)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 374 | 374
Months | 31.38 [26.18 to 36.80] | 29.47 [23.49 to 34.30]
Statistical Analysis 1: Comparison: E-Ld Cohort vs Ld Cohort; Test type: Superiority; p = 0.4358, Stratified Log Rank
Statistical Analysis 2: Comparison: E-Ld Cohort vs Ld Cohort; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95.71% CI 2-sided [0.77 to 1.12] — E-Ld/Ld. Calculated using Cox proportional hazards modeling

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with objective response among all randomized subjects. Participants with an objective response are those participants experiencing a partial response (PR) or better, based on Independent Review Committee (IRC) assessment, as per EBMT criteria.
Time Frame: From randomization to primary completion date (approximately 8 years)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 374 | 374
Percent of Participants | 82.9 [78.7 to 86.6] | 79.4 [75.0 to 83.4]
Statistical Analysis 1: Comparison: E-Ld Cohort vs Ld Cohort; Test type: Superiority; p = 0.2232, CMH ESTIMATE OF COMMON ODDS RATIO; CMH ESTIMATE OF COMMON ODDS RATIO = 1.26, 95% CI 2-sided [0.87 to 1.82]

3. Secondary Outcome: Overall Survival (OS)
Description: Survival is defined as the time from randomization to the date of death. A participant who did not die had his or her survival duration censored at the date of last contact ('last known date alive").
Time Frame: From randomization to the date of death (up to 8 years)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 374 | 374
Months | 60.42 [52.76 to 67.35] | 57.56 [48.95 to 66.56]
Statistical Analysis 1: Comparison: E-Ld Cohort vs Ld Cohort; Test type: Superiority; p = 0.8932, Stratified log rank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.19] — Stratified by stage of disease (International Staging System 1 - 2 vs 3), age (<75 years old vs >= 75 years old) and ECOG performance status (0 vs 1 - 2) at randomization

4. Secondary Outcome: Mean Change From Baseline of Pain Severity Score and Pain Interference Score
Description: Pain severity (sensory dimension) and pain interference (reactive dimension, assessing the degree to which pain interferes with function) are measured using the Brief Pain Inventory- Short Form (BPI-SF).
  BPI-SF numeric rating scale goes from 0 (No pain) to 10 (Pain as bad as you can imagine).
Time Frame: From Baseline to End of Treatment (approximately 8 years)
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Rating score
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 374 | 374
Rating score
  Pain Severity | 0.02 (2.645) | -0.25 (2.721)
  Pain Interference | 0.33 (3.077) | -0.18 (3.082)

5. Secondary Outcome: Progression Free Survival (PFS) Rate at Specific Time-points
Description: PFS rate is defined as the percentage of participants experiencing PFS at the defined time-points.
Time Frame: From randomization to the specified time-point (up to 5 years)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 374 | 374
Percent of participants
  1 year | 0.77 [0.72 to 0.81] | 0.76 [0.71 to 0.80]
  2 year | 0.59 [0.53 to 0.64] | 0.55 [0.49 to 0.60]
  3 year | 0.46 [0.40 to 0.51] | 0.41 [0.35 to 0.46]
  4 year | 0.36 [0.31 to 0.41] | 0.33 [0.28 to 0.38]
  5 year | 0.26 [0.21 to 0.32] | 0.25 [0.20 to 0.30]
Statistical Analysis 1: Comparison: E-Ld Cohort vs Ld Cohort; Test type: Superiority; p = 0.4358, Hazard Ratio; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.78 to 1.12]

ADVERSE EVENTS:
Time Frame: All-cause mortality: from first patient first visit to study completion: approximately up to 10 years and 1 month. Serious and non serious AEs: From first dose to 60 days after last dose (on average 34 months up to approximately 113 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication"
Arm/Group | E-Ld Cohort | Ld Cohort
All-Cause Mortality (participants affected / at risk) | 240/374 | 232/374
Serious Adverse Events (participants affected / at risk) | 293/371 | 279/371
Other Adverse Events (participants affected / at risk) | 364/371 | 365/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-Ld Cohort (N=371) | Ld Cohort (N=371)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 12 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 3
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0
Plasmacytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 7 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve calcification (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 22 | 12
Atrial flutter (Cardiac disorders) | 4 | 3
Atrial tachycardia (Cardiac disorders) | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 7 | 6
Cardiac failure (Cardiac disorders) | 13 | 7
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 4
Cardiac septal hypertrophy (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 2 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 6 | 5
Myocardial ischaemia (Cardiac disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 3 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Systolic dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Blindness transient (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 10 | 9
Cataract cortical (Eye disorders) | 1 | 0
Epiretinal membrane (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anorectal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 10
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 2
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oroantral fistula (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 6
Chest pain (General disorders) | 2 | 4
Complication associated with device (General disorders) | 1 | 0
Death (General disorders) | 2 | 3
Disease progression (General disorders) | 8 | 5
Fat necrosis (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 3 | 5
Inflammation (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 3
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 4
Pain (General disorders) | 1 | 3
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 19 | 7
Sudden cardiac death (General disorders) | 1 | 1
Sudden death (General disorders) | 2 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial prostatitis (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 18 | 6
Bursitis infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 9 | 8
Cellulitis orbital (Infections and infestations) | 1 | 1
Central nervous system infection (Infections and infestations) | 1 | 0
Clostridial sepsis (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 1
Dacryocystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 5 | 3
Erysipelas (Infections and infestations) | 2 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Febrile infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 8 | 2
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 4 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 7 | 6
Intervertebral discitis (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 1
Leishmaniasis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 9 | 8
Meningitis listeria (Infections and infestations) | 1 | 1
Metapneumovirus bronchiolitis (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Plague (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 60 | 48
Pneumonia aspiration (Infections and infestations) | 5 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 2 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 2
Pyoderma (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 8 | 3
Sepsis (Infections and infestations) | 15 | 6
Septic shock (Infections and infestations) | 4 | 6
Staphylococcal infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 15 | 11
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 5 | 5
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 1
Whipple's disease (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Combined tibia-fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 4 | 8
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 5 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 4
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 4
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 3
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 2 | 2
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0
Influenza B virus test positive (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0
Respirovirus test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Viral test positive (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Alcohol intolerance (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 5
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 10
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Refractory anaemia with ringed sideroblasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 7
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 7
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 3
Cerebral infarction (Nervous system disorders) | 2 | 2
Cerebral ischaemia (Nervous system disorders) | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 8 | 7
Cognitive disorder (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 4 | 1
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 7 | 5
Transient aphasia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 6 | 4
Device dislocation (Product Issues) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 5 | 5
Delirium (Psychiatric disorders) | 2 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 20 | 20
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Myeloma cast nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 10 | 7
Renal impairment (Renal and urinary disorders) | 1 | 3
Renal injury (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 9 | 10
Embolism (Vascular disorders) | 3 | 0
Embolism venous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 7 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-Ld Cohort (N=371) | Ld Cohort (N=371)
Anaemia (Blood and lymphatic system disorders) | 153 | 160
Leukopenia (Blood and lymphatic system disorders) | 23 | 37
Neutropenia (Blood and lymphatic system disorders) | 93 | 117
Thrombocytopenia (Blood and lymphatic system disorders) | 66 | 69
Atrial fibrillation (Cardiac disorders) | 28 | 25
Cataract (Eye disorders) | 61 | 56
Vision blurred (Eye disorders) | 28 | 28
Abdominal pain (Gastrointestinal disorders) | 50 | 51
Abdominal pain upper (Gastrointestinal disorders) | 33 | 29
Constipation (Gastrointestinal disorders) | 142 | 144
Diarrhoea (Gastrointestinal disorders) | 192 | 180
Dry mouth (Gastrointestinal disorders) | 28 | 26
Dyspepsia (Gastrointestinal disorders) | 43 | 32
Haemorrhoids (Gastrointestinal disorders) | 10 | 19
Nausea (Gastrointestinal disorders) | 117 | 108
Toothache (Gastrointestinal disorders) | 24 | 15
Vomiting (Gastrointestinal disorders) | 69 | 50
Asthenia (General disorders) | 88 | 73
Chest pain (General disorders) | 24 | 32
Chills (General disorders) | 35 | 9
Fatigue (General disorders) | 183 | 188
Influenza like illness (General disorders) | 40 | 28
Mucosal inflammation (General disorders) | 21 | 8
Non-cardiac chest pain (General disorders) | 20 | 19
Oedema (General disorders) | 17 | 19
Oedema peripheral (General disorders) | 163 | 182
Pain (General disorders) | 24 | 19
Peripheral swelling (General disorders) | 24 | 24
Pyrexia (General disorders) | 111 | 77
Bronchitis (Infections and infestations) | 46 | 52
Cellulitis (Infections and infestations) | 21 | 26
Cystitis (Infections and infestations) | 13 | 20
Herpes zoster (Infections and infestations) | 23 | 18
Influenza (Infections and infestations) | 14 | 20
Nasopharyngitis (Infections and infestations) | 60 | 62
Oral herpes (Infections and infestations) | 23 | 11
Pneumonia (Infections and infestations) | 33 | 23
Respiratory tract infection (Infections and infestations) | 38 | 34
Sinusitis (Infections and infestations) | 23 | 17
Upper respiratory tract infection (Infections and infestations) | 82 | 84
Urinary tract infection (Infections and infestations) | 58 | 56
Contusion (Injury, poisoning and procedural complications) | 47 | 53
Fall (Injury, poisoning and procedural complications) | 33 | 32
Skin abrasion (Injury, poisoning and procedural complications) | 24 | 13
Skin laceration (Injury, poisoning and procedural complications) | 19 | 23
Alanine aminotransferase increased (Investigations) | 18 | 27
Aspartate aminotransferase increased (Investigations) | 17 | 21
Blood creatinine increased (Investigations) | 56 | 72
Glomerular filtration rate decreased (Investigations) | 20 | 17
Neutrophil count decreased (Investigations) | 11 | 28
Platelet count decreased (Investigations) | 12 | 20
Weight decreased (Investigations) | 79 | 66
Decreased appetite (Metabolism and nutrition disorders) | 100 | 86
Dehydration (Metabolism and nutrition disorders) | 25 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 120 | 69
Hypoalbuminaemia (Metabolism and nutrition disorders) | 24 | 21
Hypocalcaemia (Metabolism and nutrition disorders) | 73 | 75
Hypokalaemia (Metabolism and nutrition disorders) | 84 | 91
Hypomagnesaemia (Metabolism and nutrition disorders) | 41 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 27 | 17
Hypophosphataemia (Metabolism and nutrition disorders) | 20 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 111 | 121
Back pain (Musculoskeletal and connective tissue disorders) | 133 | 136
Bone pain (Musculoskeletal and connective tissue disorders) | 58 | 57
Joint swelling (Musculoskeletal and connective tissue disorders) | 19 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 84 | 83
Muscular weakness (Musculoskeletal and connective tissue disorders) | 45 | 52
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 49 | 50
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 28 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 30 | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 76 | 78
Pain in jaw (Musculoskeletal and connective tissue disorders) | 19 | 12
Spinal pain (Musculoskeletal and connective tissue disorders) | 15 | 23
Dizziness (Nervous system disorders) | 84 | 68
Dysgeusia (Nervous system disorders) | 26 | 13
Headache (Nervous system disorders) | 61 | 50
Hypoaesthesia (Nervous system disorders) | 24 | 25
Memory impairment (Nervous system disorders) | 27 | 15
Neuropathy peripheral (Nervous system disorders) | 41 | 48
Paraesthesia (Nervous system disorders) | 40 | 45
Peripheral sensory neuropathy (Nervous system disorders) | 57 | 59
Syncope (Nervous system disorders) | 18 | 20
Taste disorder (Nervous system disorders) | 24 | 27
Tremor (Nervous system disorders) | 61 | 55
Agitation (Psychiatric disorders) | 21 | 17
Anxiety (Psychiatric disorders) | 44 | 28
Confusional state (Psychiatric disorders) | 37 | 32
Depression (Psychiatric disorders) | 42 | 31
Insomnia (Psychiatric disorders) | 98 | 96
Mood altered (Psychiatric disorders) | 25 | 17
Dysuria (Renal and urinary disorders) | 16 | 19
Pollakiuria (Renal and urinary disorders) | 14 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 120 | 106
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 45 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 87 | 93
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 24 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 26 | 26
Productive cough (Respiratory, thoracic and mediastinal disorders) | 33 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 22
Erythema (Skin and subcutaneous tissue disorders) | 19 | 21
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 36 | 26
Night sweats (Skin and subcutaneous tissue disorders) | 24 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 39 | 43
Rash (Skin and subcutaneous tissue disorders) | 90 | 86
Skin lesion (Skin and subcutaneous tissue disorders) | 19 | 17
Deep vein thrombosis (Vascular disorders) | 20 | 26
Flushing (Vascular disorders) | 19 | 17
Hypertension (Vascular disorders) | 54 | 44
Hypotension (Vascular disorders) | 63 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT01335399/Prot_001.pdf
  • Statistical Analysis Plan (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT01335399/SAP_000.pdf